CLINICAL TRIAL: NCT07222397
Title: Evaluation of the 2910 nm Erbium-Doped Fluoride Fiber Glass Laser for the Treatment of Advanced Perioral Lines and Wrinkles
Brief Title: 2910 nm Erbium-Doped Fluoride Fiber Glass Laser for the Treatment of Advanced Perioral Lines and Wrinkles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FA Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC 26-2025
Record Dates: First submitted 2025-02-21; First posted 2025-10-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Photodamaged Skin; Rhytids; Lines Skin; Wrinkles and Rhytides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Part 2 Clinical Study Procedure (Experimental): UltraClear 2,910nm mid-infrared laser using both superficial epidermal ablation and deep ablative and coagulative capabilities in the dermis for rejuvenation addressing perioral lines and wrinkles.
  Interventions: Device: Laser Resurfacing

INTERVENTIONS:
Device: Laser Resurfacing — Enrolled participants will be treated with the UltraClear 2,910nm mid-infrared laser using both superficial epidermal ablation and deep ablative and coagulative capabilities in the dermis for rejuvenation with a specific focus on perioral lines and wrinkles.
  Other Names: Ablative Fractional Laser Resurfacing; 2910 nm mid-infrared fiber laser

SUMMARY:
The primary objective is to assess the efficacy, safety and satisfaction associated with the resurfacing treatment of perioral lines and wrinkles with the 2,910 nm mid-infrared Fiber Laser (UltraClear, Acclaro Medical) using both superficial epidermis ablation capabilities and the deep ablative and coagulative capabilities into the dermis for rejuvenation.

Participants will receive up to two treatments spaced 6-8 weeks apart, followed by a 1-month and 3-month follow-up visit during which the device will be evaluated for its effectiveness defined as improvement addressing perioral lines and wrinkles utilizing multiple scales completed by the investigator and blinded Independent Photographic Reviewers (IPRs). Additionally, safety, subjective overall aesthetic improvement and satisfaction will be monitored and tracked.

ELIGIBILITY:
Inclusion Criteria:

1. Fitzpatrick skin type I-IV.
2. Male or female.
3. Subjects must be between 50 and 80 years of age.
4. Subjects must have the ability to receive up to two full face resurfacing laser treatment with specific focus on advanced perioral lines and wrinkles.
5. Subjects must read, understand, and sign the Informed Consent Form.
6. Subjects must be willing and able to comply with all follow-up visit requirements.
7. Subjects must agree to refrain from using cosmeceutical agents or topical agents during the study, except as directed by study investigator.
8. Subjects must be rated as Class II or Class III based on the Fitzpatrick Wrinkling and Degree of Elastosis Scale (FWS).
9. Subject identified as an appropriate candidate for study treatment based on principal investigator's opinion.
10. Subjects of childbearing potential have been on an acceptable form of contraception for 30 days prior to enrollment and agree to continue using throughout the course of the study.

Exclusion Criteria:

1. Subjects must not have active localized or systemic infections.
2. Subjects must not have a compromised ability for wound healing, such as: malnutrition, steroid use, history of collagen vascular disease (e.g., lupus, scleroderma, history of keloid scar formation), atrophic dermatitis or immunologic abnormalities such as vitiligo.
3. Subjects must not have had treatments with 5FU, diclofenac, imiquimod, steroids, retinoids, or PDT within 1-month prior to enrollment.
4. Subjects must not currently be taking Accutane or have taken Accutane within the last 1-month.
5. Subjects must not have a known allergy to lidocaine or epinephrine, topical or injectable products containing lidocaine or any numbing medications.
6. Subjects must not have had previous surgery and/or fat transfer in the treatment area within the last 6-months.
7. Subject must not have had injectable soft tissue fillers within the last 12 months in the treatment area.
8. Subject must not have had Poly-L-Lactic acid (PLLA) fillers within the last 2 years in the treatment area.
9. Subject must not have had permanent filler i.e., Polymethylmethacrylate (PMMA) in the treatment area.
10. Subjects must not have had neurotoxins within the last 3-months in the treatment area.
11. Subject must not have a personal history of any facial threads i.e., PDO (Polydioxanone), PLLA (Polylactic acid), PCL (Polycaprolactone) in the treatment area within the last 12 months.
12. Subject must not have had a pulse dye or vascular laser, non-ablative laser, microneedling, or energy-based device treatment in the treatment area within the last 3 months.
13. Subject must not have had an ablative laser treatment in the treatment area within the last 6 months.
14. Subjects must not have a personal history of malignant melanoma, keloid scars, generalized psoriasis or systemic diseases that would preclude the use of topical anesthesia.
15. Subject must not have active sunburn or excessively tanned skin.
16. Subjects must not be pregnant or breastfeeding, think they may be pregnant or are trying to get pregnant during the study.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in Fitzpatrick Wrinkling and Degree of Elastosis Scale (FWS) | From enrollment to the final follow-up visit (3-months following final treatment)
  Changes in perioral lines and wrinkles utilizing the Fitzpatrick Wrinkling and Degree of Elastosis Scale (FWS).
  A change of one point is considered a statistically significant change on a scale of 1-9, with one being the least noticeable wrinkles and nine being the deepest and most noticeable wrinkles.
  1 - 3 Fine wrinkles 4 - 6 Fine to moderate depth wrinkles, moderate number of lines 7 - 9 Fine to deep wrinkles, numerous lines, with or without redundant skin folds
Percentage of Treatment Responders | From enrollment to the final follow-up visit (3-months following final treatment)
  o Comparison of the proportion of subjects (i.e., percentage of treatment responders) correctly identified by at least two out of three blinded Independent Photographic Reviewers (IPR).
Change in Physician Global Aesthetic Improvement Scale (PGAIS) | From enrollment to the final follow-up visit (3-months following final treatment)
  Defined as a change in perioral lines and wrinkles utilizing the Physician Global Aesthetic Improvement Scale (PGAIS).
  The PGAIS is a five-point scale used by physicians to objectively rate the aesthetic outcome of a treatment by comparing a patient's pre-treatment and post-treatment appearance.
  The scoring is numerical (1-5), with a score of 3, 4, or 5 points being considered significant.
  1. - Worse: The patient's aesthetic appearance has deteriorated compared to baseline
  2. - No Change: There is no noticeable difference from the pre-treatment state.
  3. - Improved: The physician notes a visible enhancement, but further treatment could still be beneficial
  4. - Much Improved: There is a marked, clear aesthetic improvement
  5. - Very Much Improved: An optimal cosmetic result has been achieved

SECONDARY OUTCOMES:
Subject Self-Reported Improvements | From enrollment to the final follow-up visit (3-months following final treatment)
  The SGAIS is a measure of aesthetic improvement relative to baseline, pre-treatment condition. A meaningful change on the Subject Global Aesthetic Improvement Scale (SGAIS) is defined as an improvement of at least one grade, indicating that the subject perceives a beneficial change in their appearance. The SGAIS is a patient-reported outcome measure (PROM) that is completed by the patient/subject to assess their own perception of aesthetic improvement following treatment.
  The scale is reported with scores of 1-5.
  1. - Worse: The subject perceives a deterioration in their appearance compared to before treatment
  2. - No Change: There is no noticeable difference from the pre-treatment state
  3. - Improved: The subject notes a visible aesthetic improvement
  4. - Much Improved: The subject notes marked and definite aesthetic improvement
  5. - Very Much Improved: The subject believes an optimal comment result has been achieved

CONTACTS AND LOCATIONS:
Overall Officials: Paul Friedman, MD, Principal Investigator — Director, Dermatology & Laser Surgery Center Clinical Assistant Professor of Dermatology, UT Medical School
Locations (1):
- Dermatology & Laser Surgery Center, Houston, Texas, United States

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT07222397/SAP_000.pdf